CLINICAL TRIAL: NCT06562894
Title: A Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate the Efficacy and Safety of SYHX1901 Tablets in the Treatment of Severe Alopecia Areata
Brief Title: Study to Evaluate Safety and Efficacy of SYHX1901 Tablets in Severe Alopecia Areata Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Collaborators: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYHX1902-006
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Severe Alopecia Areata
Keywords: plaque psoriasis
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SYHX1901 dose 1 (Experimental)
  Interventions: Drug: SYHX1901
- SYHX1901 dose 2 (Experimental)
  Interventions: Drug: SYHX1901
- SYHX1901 dose 3 (Experimental)
  Interventions: Drug: SYHX1901
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYHX1901 — Administered orally, once daily (QD)
  Arms: SYHX1901 dose 1; SYHX1901 dose 2; SYHX1901 dose 3
Drug: Placebo — Administered orally, once daily (QD)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of different doses of SYHX1901 tablets in the treatment of severe alopecia areata.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled phase II study to evaluate the efficacy and safety of two different doses of SYHX1901 tablets compared with placebo in the treatment of severe alopecia areata. The total duration of the study will be 56 60 weeks which will be comprised of: a screening period (4 weeks); a core treatment period (24 weeks),a extended treatment period（28 weeks）and a follow-up assessment period (4 weeks). Eligible subjects will be randomly assigned to SYHX1901 dose 1 , dose 2，dose 3 or placebo group at a 1:2:2:1 ratio for continuous oral administration for 24 weeks, then placebo group will receive SYHX1901 at dose 3 for 28 weeks, the SYHX1901 dose 1, dose 2，dose 3 group will remain the same dose for 28 weeks. The SALT（Severity of AlLopecia Tool） score will be a stratification factor. Subjects will be monitored for the safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent;
2. Subjects aged ≥18 to ≤ 65 years;
3. Clinical diagnosis of alopecia areata,with at least 50% scalp hair loss，as defined by a SALT score ≥50 at screening and baseline visit;
4. The current episode of hair loss was less than 10 years ago, and there was no evidence of spontaneous hair regrowth within 6 months before screening (the overall duration of alopecia areata more than 10 years could be included);
5. Subjects must be volunteer and be able to understand informed consent Forms;
6. Subjects and their partners should voluntarily take contraceptive measures considered effective by the investigator during the study period and for at least 28 days after the study;

Exclusion Criteria:

1. Participants who have received hair implants;
2. Alopecia caused by other reasons;
3. Other active scalp or systemic diseases that may cause severe alopecia or affect the clinical evaluation of alopecia areata;
4. Participants who have shaved their heads;
5. Participants who have a clinically significant (as assessed by the investigator) abnormality in TSH or free T4 at screening and who were deemed by the investigator to be ineligible for the study;
6. Participants who wore stick-on wigs and refused to stop wearing them during the study;
7. Bacterial, fungal, or viral infection requiring hospitalization/intravenous treatment within 4 weeks before the first dose of study drug or requiring oral treatment within 2 weeks before the first dose of study drug;
8. Have any chronic infection that requires systemic anti-infective therapy;
9. Have received a live vaccine within 60 days before the first dose of the study drug or plan to receive a live vaccine between the middle of the study and 60 days after the end of the study;
10. History of severe herpes zoster or sever herpes simplex infection;
11. HBV-related tests are abnormal at screening;
12. HCV antibody positive and HCV RNA positive at screening;
13. Human immunodeficiency virus antibody positive or treponema pallidum antibody positive;
14. Any known or suspected condition of congenital or acquired immunodeficiency;
15. Previous or current active tuberculosis infection or latent tuberculosis infection (LTBI) deemed by the investigator/specialist to require treatment;
16. Major surgery within 8 weeks prior to first dose of the study drug or planned surgery during the study;
17. Organ transplantation (except corneal transplantation more than 3 months before the initiation of the investigational drug);
18. Symptoms or signs of progressive or uncontrolled kidney, liver, blood, gastrointestinal, endocrine, lung, heart, neurological, psychiatric, or brain disease, or with other chronic diseases that the investigator has determined are not suitable for participation in this clinical trial;
19. History of malignancy or lymphoproliferative disease;
20. Uncontrolled hypertension, systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg after systemic treatment;
21. Having unstable cardiovascular disease defined as presence of a clinical cardiovascular event in the last 3 months or hospitalized for heart disease within the last 3 months; or NYHA≥grade 3, or abnormal ECG suggesting clinically significant and assessed by the investigator as carrying unforeseen risks;
22. Patients with a history of arterial or venous thrombosis or high risk factors for thrombosis within 6 months before the first dose of study drug;
23. Combined with active lipid-lowering drugs but poorly controlled hyperlipidemia: total cholesterol (TC)≥ 6.2mmol/L or low-density lipoprotein cholesterol (LDL-C)≥3.4mmol/L; or familial hypercholesterolemia (FH);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-05-26 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-11-17 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with Alopecia Severity Score Tool (SALT) score < or = 20% | Week 24
  Percentage of subjects achieving a SALT score < or = 20% at week 24

IPD SHARING:
Plan to Share IPD: No